CLINICAL TRIAL: NCT04221503
Title: A Phase II Study Evaluating the Efficacy and Safety of Niraparib and Tumor-Treating Fields in Recurrent Glioblastoma
Brief Title: Niraparib/TTFields in GBM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Tesaro, Inc. (Industry); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03319
Record Dates: First submitted 2019-12-17; First posted 2020-01-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma | interventions — niraparib; Transurethral Resection of Bladder

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cohort A (Experimental): Cohort A is for subjects with recurrent glioblastoma who do not have clinical indication for surgical resection of the recurrent tumor. Subjects in Cohort A will initiate and continue TTFields therapy for 5-7 days prior to starting niraparib.
  Interventions: Drug: Niraparib; Device: Optune
- Cohort B (Active Comparator): Cohort B is for subjects with recurrent glioblastoma who have a clinical indication for surgical resection of the recurrent tumor. Subjects in Cohort B will receive TTFields for 5-7 days prior to planned surgical resection, undergo surgical resection, resume TTFields postoperatively, and initiate niraparib 5- 7 days after starting TTFields postoperatively.
  Interventions: Drug: Niraparib; Device: Optune; Procedure: Planned surgical resection

INTERVENTIONS:
Drug: Niraparib — Niraparib ([3S]-3-[4-{7-(aminocarbonyl)-2H-indazol-2-yl} phenyl] piperidine [tosylate monohydrate salt]) is an orally available, potent, highly selective poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) -1 and -2 inhibitor. The niraparib drug product is provided as 100-mg capsules filled with a dry blend of niraparib tosylate monohydrate, lactose monohydrate, and magnesium stearate in a hard gelatin capsule.
  Other Names: ZEJULA
Device: Optune — Optune, which is manufactured by Novocure, is a portable battery or power supply operated device which produces alternating electrical fields, called tumor treatment fields ("TTFields") within the human body. TTFields are applied to the patient by electrically-insulated surface transducer arrays. TTFields disrupt the rapid cell division exhibited by cancer cells.
  Other Names: Tumor Treatment Fields (TTFields)
Procedure: Planned surgical resection — Surgery of supratentorial glioblastoma (GBM).
  Other Names: Tumor Resection
  Arms: Cohort B

SUMMARY:
Evaluating the efficacy and safety of niraparib and Tumor-Treating Fields (TTFields) in recurrent glioblastoma (GBM).

DETAILED DESCRIPTION:
Tumor-treating fields (TTFields) causes downregulation of BRCA1 signaling and reduced deoxyribonucleic acid (DNA) double-strand break repair capacity. Tumors that are deficient in the homologous recombination DNA damage repair pathway are highly sensitive to blockade of the repair of single strand DNA breaks via poly-ADP ribose polymerase (PARP) inhibition. This is a study of niraparib, a PARP inhibitor, in combination with tumor-treating fields for recurrent glioblastoma. We hypothesize that tumor-treating fields will induce a state of "BRCAness" in the glioma tumor cells, thus sensitizing them to PARP inhibition and resulting in tumor cell death.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or molecularly (per c-IMPACT NOW criteria) proven diagnosis of glioblastoma which is recurrent following radiation therapy (prior dose must have been between 40 and 75 Gy).
* Tumor O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation status must be available from any prior GBM tumor specimen.
* Patients must have measurable contrast-enhancing disease (defined by at least 1cm x 1cm) by magnetic resonance imaging (MRI) imaging within 28 days of starting study treatment.
* Patients may have had treatment for an unlimited number of prior relapses.
* Patients must have recovered from severe toxicity of prior therapy.
* Patients must be able to swallow oral medications.
* Karnofsky performance status >= 60.
* Life expectancy >3 months.
* Adequate hematologic parameters.
* Adequate hepatic function within 7 days prior to start of study treatment.
* Adequate renal function within 7 days prior to start of study treatment.
* Reproductive Status
* Women - negative serum or urine pregnancy test
* Men and Women - must agree to an adequate method to avoid pregnancy
* Participant must agree to not donate blood during the study or for 90 days after the last dose of niraparib.
* Participant must, in the opinion of the Investigator, be able to comply with study procedures, including use of the Optune device.
* Cohort B (surgical) patients only: patients must be undergoing surgery that is clinically indicated as determined by their care providers.
* Cohort B (surgical) patients only: patients must have a tumor tissue form indicating availability of archived tissue from a previous surgery for glioblastoma.
* Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent (or have legally authorized representative sign on patient's behalf if patient physically unable to sign consent due to neurologic deficit).

Exclusion Criteria:

* Age < 22 years.
* Prior treatment with tumor-treating fields therapy (Optune) within the past 6 months.
* Prior treatment with a PARP inhibitor.
* Known history or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML).
* Patients with infratentorial tumor.
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
* Implanted pacemaker, defibrillator or deep brain stimulator, other implanted electronic devices in the brain. Non-programmable shunts are allowed. Patients with a programmable shunt are excluded.
* Skull defects.
* Known hypersensitivity to conductive hydrogels or known hypersensitivity to niraparib components or excipients.
* Patients with gastrointestinal disorders or abnormalities that would interfere with absorption of study treatment.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Participant must not be simultaneously enrolled in any interventional clinical trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Disease control, defined as achievement of either CR, PR, or SD, as defined by modified Response Assessment in Neuro-Oncology (mRANO) criteria. | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Complete response (CR) is seen as the disappearance of all enhancing measurable and non-measurable disease sustained for at least 4 weeks.
  Partial response (PR) is ≥50% decrease in sum of products of perpendicular diameters or ≥65% decrease in total volume of all measurable enhancing lesions compared with baseline, sustained for at least 4 weeks.
  Stable disease (SD), must be present on two consecutive MRI scans, with the 2nd/confirmatory MRI performed at least 16 weeks after starting treatment.

SECONDARY OUTCOMES:
Number of AEs (Adverse Events) | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, all events will be recorded from the time a subject has signed the informed consent form.
Duration of disease control. | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Achieving a confirmed best response to treatment of stable disease (SD), partial response (PR), or complete response (CR).
Objective radiographic response (ORR) | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  ORR is defined by mRANO criteria, and duration of response.
Progression-free survival (PFS) | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Progression-free survival (PFS) is defined as the time from date of enrollment until the earliest date of disease progression (as determined by mRANO criteria) or death due to any cause.
Overall survival (OS) | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Overall survival (OS) is defined as the time from date of enrollment until death from any cause.

OTHER OUTCOMES:
Objective response rate (ORR) associations. | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Association between pre-treatment tumor genomics, transcriptomics, proteomics, and prior bevacizumab use and ORR.
Progression-free survival (PFS) associations | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Association between pre-treatment tumor genomics, transcriptomics, proteomics, and prior bevacizumab use and PFS.
Overall survival (OS) associations | When termination of the study or 5 years after removal from protocol therapy, whichever occurs first.
  Association between pre-treatment tumor genomics, transcriptomics, proteomics, and prior bevacizumab use and OS.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No